CLINICAL TRIAL: NCT03705390
Title: A Phase II Pilot Single-arm Safety and Tolerability Study of ILB® in Patients With Motor Neurone Disease (MND)/ Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Safety and Tolerability Study of ILB® in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study initially suspended due to COVID-19 Pandemic- treatment stopped - never reopened to recruitment..
Sponsor: University of Birmingham (Other)
Collaborators: TikoMed AB (Industry); University Hospital Birmingham (Other); Neuregenix Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_17-250
Record Dates: First submitted 2018-09-11; First posted 2018-10-15 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: ILB; Amyotrophic Lateral Sclerosis; Motor Neuron Disease; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ILB® Arm (Experimental): ILB® subcutaneous injection at a dose of 2mg/kg once per week for up to a maximum of 48 weeks
  Interventions: Drug: ILB®

INTERVENTIONS:
Drug: ILB® — Administration will be weekly subcutaneous injections at a dose of 2mg/kg once per week for up to a maximum of 48 weeks
  Other Names: DSSS5; TM-500; TM-700; LMW-DS; IBsolvMIR

SUMMARY:
This is a phase II study to determine the safety and tolerability of ILB®, a type of low molecular weight dextran sulfate, in patients with Motor Neurone Disease (MND)/ Amyotrophic Lateral Sclerosis (ALS)

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) belongs to a wider group of disorders known as motor neuron diseases and mainly involves the nerve cells (neurons) in the body. Voluntary muscles produce movements like chewing, walking and talking. ALS is caused by gradual deterioration (degeneration) and death of these motor neurons. The disease is progressive, meaning the symptoms get worse over time and most people with ALS die from respiratory failure, usually within 3 to 5 years from when the symptoms first appear. Currently there is no cure for ALS and no effective treatment to halt or reverse the progression of the disease (National Institute of Neurological Disorders and Stroke, Fact Sheet).

The aim of this study is to explore the safety and acceptability of a type of low molecular weight dextran sulfate called ILB®.

The investigators will invite 15 patients to take part from a single centre in the United Kingdom (UK). Participants will be closely monitored for any side-effects; for changes in ALS symptoms and on quality of life during and after the study.

The trial period for patient participation is maximum 56 weeks (12 months), ILB® injections will be administered once weekly for up to a maximum of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years and who have provided written informed consent to participate in the study
2. Prior to trial entry patients will have a definite diagnosis of ALS according to El Escorial Criteria. All patients will demonstrate either:

   * presence of Upper Motor Neuron (UMN) (increased tone, brisk reflexes) as well as Lower Motor Neuron (LMN) (weakness,
   * wasting and fasciculation) signs in the bulbar region and at least two of the other spinal regions (cervical, thoracic or lumbosacral) or
   * presence of UMN and LMN signs in all three spinal regions (cervical, thoracic or lumbosacral)
3. Electrophysiological tests (Electromyography (EMG) / Nerve Conduction Study (NCS)) that supports the diagnosis of Motor Neurone Disease (MND) and to exclude mimic disorders
4. Forced Vital Capacity (FVC) ≥50% of predicted value for gender, height and age at screening and a mean Sniff Nasal Inspiratory Pressure (SNIP) ≥50% of predicted value for age
5. Adequate haematological function (Hb≥10g/dl absolute neutrophil count ≥1.5x109/L and a platelet count ≥60 x109/L
6. International Normalised Ratio (INR) ≤ 1.5, Activated Partial Thromboplastin Time (aPTT) 30 - 40 seconds, Prothrombin Time (PT) 11-13.5 seconds
7. Patient willing and able to comply with schedule visits, treatment plan and other study procedures.
8. Patients taking Riluzole must have discontinued treatment ≥28 days prior to study entry (and following consent to take part in the study)
9. Women Of Child Bearing Potential (WOCBP) who agree to use highly effective means of contraception (as defined in the Heads of Medicines Agencies_Clinical Trials Facilitation Group (HMA_CTFG) guideline (see Appendix 8) and in combination with a barrier contraception method (condom, diaphragm or cap) for the entirety of the study

Exclusion Criteria:

1. Patients classified as either probable or possible ALS according to El Escorial Criteria.
2. Subjects in whom other causes of neuromuscular weakness have not been excluded
3. Assisted ventilation of any type within 3 months before the screening visit or at screening
4. Patients requiring Radiologically Inserted Gastrostomy (RIG) or Percutaneous Endoscopic Gastroscopy (PEG) feeding
5. Involvement in any other interventional study involving use of another Investigational Medicinal Product (IMP) or biological product, within 3 months of screening
6. Any use of antioxidants, edaravone, tirasemtiv or CK-2127107 within 1 month before the screening visit
7. Any botulinum toxin use within 3 months before the screening visit.
8. Any form of stem cell or gene therapy for the treatment of amyotrophic lateral sclerosis (ALS)
9. Neuroimaging of brain and cervical spine with Magnetic Resonance imaging (MRI) indicating compressive myelopathy as an alternate diagnosis
10. Laboratory examinations including Acetylcholine receptor (AChR) antibodies and Muscle Specific Kinase (MuSK) antibodies to exclude Bulbar onset Myasthenia gravis from Bulbar onset Motor neuron disease as an alternate diagnosis and Antinuclear Antibodies (ANA), Anti-neutrophil cytoplasmic antibodies (ANCA), Extractable Nuclear Antigen (ENA) antibodies, Creatine Kinase (CK), electrophoresis and immunoglobulin indicating an alternate diagnosis for muscle disease like Myositis
11. Abnormal liver function defined as Aspartate Transaminase (AST) and/or Alanine Transaminase (ALT) >3 times upper limit of normal
12. Any head trauma, intracranial or spinal surgery within 3 months of trial entry
13. Patients who have had recurrent falls will be excluded to reduce the risk of intracerebral haemorrhage with this IMP
14. Current use of an anticoagulant e.g Warfarin, Aspirin, Clopidogrel, any novel anticoagulants (NOAC)s or low molecular weight subcutaneous heparin
15. Uncontrolled severe hypertension defined as systolic blood pressure (SBP) ≥ 220 mmHg or diastolic blood pressure (DBP) ≥120 mmHg
16. Current or previous history of heparin-induced thrombocytopenia
17. Active peptic ulcer disease
18. Known hypersensitivity to sulphur
19. Severe liver insufficiency
20. Patients with evidence of major psychiatric illness, significant cognitive impairment or clinically evident dementia that may interfere with the patients' ability to comply with study procedures
21. Pulmonary illness (e.g asthma or Chronic Obstructive Pulmonary Disease (COPD)) requiring regular treatment
22. Patient judged to be actively suicidal by the investigator during 3 months before the screening visit
23. Subjects with a diagnosis of another neurodegenerative disease (e.g. Parkinson's disease, Alzheimer's disease and Frontotemporal dementia)
24. Pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkataramanan Srinivasan, MRCP, MRCP, Principal Investigator — University of Birmingham
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srinivasan V, Homer V, Barton D, Clutterbuck-James A, Jenkins S, Potter C, Brock K, Logan A, Smith D, Bruce L, Nagy Z, Bach SP. A low molecular weight dextran sulphate, ILB(R), for the treatment of amyotrophic lateral sclerosis (ALS): An open-label, single-arm, single-centre, phase II trial. PLoS One. 2024 Jul 11;19(7):e0291285. doi: 10.1371/journal.pone.0291285. eCollection 2024. PMID 38990927

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Weekly dosing for 10 weeks (in the first instance) during out-patient visits at site. Dosing beyond 10 weeks (initially to 24 weeks and then up to a maximum of up to 48 weeks) was dependent upon a formal review of the patient's eligibility, their wishes and the most suitable treatment options.
  Following suspension of the trial due to the COVID-19 pandemic, patients were asked to re-consent for an additional single point long-term remote follow up visit in Quarter 1 of 2021 via video call.
Period: 10 Week Initial Treatment Period
Arm/Group | ILB® Arm
Started | 11
Completed | 9
Not Completed | 2
Not completed — Trial suspended prior to completion | 2
Period: Treatment Extension
Arm/Group | ILB® Arm
Started | 9
Completed | 8 (1 participant declined)
Not Completed | 1
Not completed — Trial closed early due to COVID-19 pandemic | 1

BASELINE CHARACTERISTICS:
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11
Time from ALS diagnosis to trial entry (months) [Mean (Standard Deviation); unit: months] | 7.27 (5.34)
Family history of motor neurone disease (n(%)) [Count of Participants; unit: Participants]
  No | 10
  Yes | 1
Family history of fronto-temporal dementia (n(%)) [Count of Participants; unit: Participants]
  No | 11
  Yes | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessed by SAEs and AEs - Measured by Incidence
Description: Measured by the number of serious adverse events (SAEs) and adverse events (AEs) using CTCAE grading v4.0.
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: Adverse events
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
Adverse events
  Serious Adverse Events | 1
  Adverse Events | 270

2. Primary Outcome: Safety Assessed by AEs - Summarised by Grade
Description: Grade refers to the severity of the AE as follows:
  Grade 1 - Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 - Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 - Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 - Life-threatening consequences; urgent intervention indicated. Grade 5 - Death related to AE.
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: number of AEs
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of AEs
  Grade 1 | 265
  Grade 2 | 4
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0

3. Primary Outcome: Safety Assessed by AEs - Summarised by Relatedness
Description: Relatedness categories: 1 = unrelated, 2 = unlikely to be related, 3 = possibly related, 4 = probably related, 5 = definitely related
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: number of AEs
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of AEs
  Unrelated | 127
  Unlikely to be related | 45
  Possibly related | 4
  Probably related | 1
  Definitely related | 93

4. Primary Outcome: Safety Assessed by SAEs - Summarised by Admitting Event Grade
Description: Grade refers to the severity of the admitting event as follows:
  Grade 1 - Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 - Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 - Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 - Life-threatening consequences; urgent intervention indicated. Grade 5 - Death related to AE.
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: number of SAEs
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of SAEs
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0

5. Primary Outcome: Safety Assessed by SAEs - Summarised by Admitting Event Relatedness
Description: as for outcome 3
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: number of SAEs
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of SAEs
  Unrelated | 1
  Unlikely to be related | 0
  Possibly related | 0
  Probably related | 0
  Definitely related | 0

6. Primary Outcome: Safety Assessed by SAEs - Summarised by Admitting Event Type
Description: Description of the main event type - primary cause of admission (body system, Adverse event term and grade)
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: number of SAEs
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of SAEs
  Musculoskeletal and connective tissue disorder - Other, specify: generalised muscle weakness | 1
  Other admitting event types | 0

7. Primary Outcome: Safety Assessed by SAEs - Summarised by Expectedness
Description: Serious Adverse Events only will be defined as expected or unexpected based on information provided in the Quick Reference Document
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Population: Expectedness of SAEs is only ascertained in the instance of the event being a Serious Adverse Reaction (SAR), therefore as the only SAE was unrelated, expectedness was not applicable
Arm/Group | ILB® Arm
Number analyzed (Participants) | 0

8. Primary Outcome: Safety Assessed by SAEs - Summarised by Sequelae
Description: Outcome of serious adverse events only: Resolved with sequelae or Resolved without sequelae
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: number of SAEs
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of SAEs
  Resolved with Sequelae | 0
  Resolved without Sequelae | 1

9. Primary Outcome: Tolerability Assessed by the Incidence of Intolerable Adverse Events
Description: An intolerable adverse event will satisfy all of the following criteria:
  1. Associated with a serious adverse event or a drug discontinuation of greater than three weeks;
  2. Grade 3, 4 or 5 in severity according to CTCAE version 4;
  3. In the opinion of the Investigator is i) definitely related or ii) probably related or iii) possibly related to the study drug treatment.
  Adverse events which are considered unrelated or probably not related will not be classed as intolerable events.
Time Frame: From informed consent up to 30 days after last administration of trial treatment
Measure: Number; unit: Number of intolerable adverse events
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
Number of intolerable adverse events | 0

10. Primary Outcome: Quantity of Study Drug Administered - Total Drug Administered
Description: Total drug administered over the study period (measured in milligrams)
Time Frame: From baseline to final treatment visit
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
mg | 4200 [1902 to 5754]

11. Primary Outcome: Quantity of Study Drug Administered - Number of Administrations
Description: Numerical count of the number of study drug injections given whilst on the trial
Time Frame: From baseline to final treatment visit
Measure: Median (Inter-Quartile Range); unit: number of drug administrations
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of drug administrations | 24 [14 to 35]

12. Primary Outcome: Quantity of Study Drug Administered - Number of Interruptions
Description: Numerical count of the number of study drug injections missed whilst on the trial
Time Frame: From baseline to final treatment visit
Measure: Median (Inter-Quartile Range); unit: number of interruptions
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of interruptions | 1 [0 to 3]

13. Primary Outcome: Quantity of Study Drug Administered - Duration of Interruptions
Description: Length of interruptions in weeks between study drug injections for those participants that experienced a treatment interruption whilst on the trial
Time Frame: From baseline to final treatment visit
Population: 6 patients experienced a treatment interruption whilst on the trial
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | ILB® Arm
Number analyzed (Participants) | 6
weeks | 1.5 [1 to 2]

14. Primary Outcome: Quantity of Study Drug Administered - Number of Discontinuations
Description: numerical count of patients who have discontinued study drug treatment
Time Frame: From baseline to final treatment visit
Measure: Number; unit: number of treatment discontinuations
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
number of treatment discontinuations | 0

15. Secondary Outcome: Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) Score Change
Description: Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R). This patient reported outcome measures the subjective well-being of patients. There are 5 scales which are calculated and scored: physical mobility, independence,eating and drinking, communication,emotional functioning. Each is scored between 0-100. An improved condition is represented by a decreasing sub-scale score. These sub scales are then averaged to make a summary index score. The range of the summary index is 0-100 and an improved condition is represented by decreasing summary index score. For each of the sub-scales and summary index. Interpretation is as follows: 0-19 Never or very rarely, 20-39 rarely experience problems, 40-59 sometimes experience problems,60-79 often experience, 80-100 problems (nearly) always or unable to do at all. The scale of the summary score is also 0-100 with analogous interpretation to the sub scales. An increase in score is a worse outcome.
Time Frame: From baseline to final treatment visit
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
score on a scale | 2.0 [0.5 to 3.0]

16. Secondary Outcome: Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) Score Change
Description: Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 . A functional rating scale including assessments of communication, mobility, dressing and respiration. the total score range is 0-40. An improved condition is represented by decreasing sub-scale score. Interpretation is as follows: 0 being the best outcome and 40 being the worst. Minimum value is 0 and Maximum value is 40 per time-point / questionnaire completion
Time Frame: From baseline to final treatment visit
Measure: Median (Inter-Quartile Range); unit: change in ALSAQ-40 score from baseline
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
change in ALSAQ-40 score from baseline
  Physical mobility | -5.0 [-15.0 to -3.8]
  Activities of daily living | -2.5 [-17.5 to 2.5]
  Eating and drinking | 0 [-12.5 to 0]
  Communication | 0 [-8.9 to 0]
  Emotional functioning | -7.5 [-18.5 to -5.0]
  Summary index score | -6.2 [-15.0 to -1.9]

17. Secondary Outcome: Urinary p75ECD Change
Description: Urinary p75 extracellular domain (p75ECD) is a biological fluid-based biomarker of ALS disease progression
Time Frame: From baseline to final treatment visit
Measure: Median (Inter-Quartile Range); unit: ng/mmol creatinine
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
ng/mmol creatinine | -0.62 [-0.98 to 0.22]

18. Secondary Outcome: Pharmacokinetics (PK; Amount of Detectable Drug) of ILB® in Plasma Following Administration
Description: This outcome measure quantifies the amount of drug detectable in the blood after administration over time
Time Frame: 0.5,1,2,2.5,3,4 and 6 hours post first ILB® administration
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | ILB® Arm
Number analyzed (Participants) | 6
μg/mL
  0.5 hours | 3.73 (1.41)
  1 hours | 4.86 (1.18)
  2 hours | 5.56 (1.45)
  2.5 hours | 5.66 (1.5)
  3.0 hours | 5.4 (1.03)
  4.0 hours | 4.76 (1.17)
  6.0 hours | 3.72 (0.76)

19. Secondary Outcome: Pharmacokinetics (PK; Tmax) Statistics of ILB® in Plasma Following Administration
Description: Tmax (the time the peak concentration occurred) was calculated to characterise the kinetic profile of ILB® in plasma post-administration
Time Frame: 0.5,1,2,2.5,3,4 and 6 hours post first ILB® administration
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ILB® Arm
Number analyzed (Participants) | 6
hours | 2.42 (0.38)

20. Secondary Outcome: Pharmacokinetics (PK; Cmax) Statistics of ILB® in Plasma Following Administration
Description: Cmax (peak concentration of ILB® in plasma post-administration) was calculated to characterise the kinetic profile of ILB® in plasma post-administration
Time Frame: 0.5,1,2,2.5,3,4 and 6 hours post first ILB® administration
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | ILB® Arm
Number analyzed (Participants) | 6
μg/mL | 6.03 (1.16)

21. Secondary Outcome: Pharmacokinetics (PK; AUC0-last) Statistics of ILB® in Plasma Following Administration
Description: AUC0-last (area under the curve time 0 (time of administration) to the last value above the limit of quantification) was calculated to characterise the kinetic profile of ILB® in plasma post-administration
Time Frame: 0.5,1,2,2.5,3,4 and 6 hours post first ILB® administration
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | ILB® Arm
Number analyzed (Participants) | 6
μg*h/mL | 27.18 (5.62)

22. Secondary Outcome: Pharmacokinetics (PK; t1/2) Statistics of ILB® in Plasma Following Administration
Description: t1/2 (terminal half-life of ILB® in plasma post-administration) was calculated to characterise the kinetic profile of ILB® in plasma post-administration
Time Frame: 0.5,1,2,2.5,3,4 and 6 hours post first ILB® administration
Population: The terminal half-life t1/2 could not be calculated for 3 out of the 6 patients as the concentration of ILB® in plasma did not drop below half its maximal value.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ILB® Arm
Number analyzed (Participants) | 3
hours | 3.74 (1.63)

23. Secondary Outcome: NfL in Plasma Change
Description: Plasma neurofilament light chain (NfL) is a blood-based biomarker for neurodegeneration
Time Frame: from baseline to final treatment visit
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | ILB® Arm
Number analyzed (Participants) | 11
ng/L | 1.5 [-3.0 to 4.5]

ADVERSE EVENTS:
Time Frame: Details of all Adverse Events (AEs) were documented and reported from the participant signing of the informed consent and included the collection of all baseline AEs. AE collection continued until 30 days after the end of treatment visit. Up to 52 weeks. The actual length of AEs collection for each participants was determined by the individual participant length of time on the study.
Description: All AEs, either observed by the Investigator or reported by the subject, were recorded by the Investigator (on an adverse event form) and evaluated. AEs were reviewed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | ILB® Arm
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ILB® Arm (N=11)
Generalised muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ILB® Arm (N=11)
Not clinically significant abnormal blood creatinine (Blood and lymphatic system disorders) | 1 (1)
Not clinically significant creatinine kinase, 286, (normal range 30-200) (Blood and lymphatic system disorders) | 1 (1)
Not clinically significant monocyte count, 0.9, (normal range 0.2 - 0.8) (Blood and lymphatic system disorders) | 1 (1)
Not clinically significant raised red cell distribution, 14.8 (normal range 11-14) (Blood and lymphatic system disorders) | 1 (1)
'Sticky' left eye (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Chesty cough (General disorders) | 1 (1)
Cold chills down left arm (General disorders) | 1 (1)
Cramps in the chest and abdomen (General disorders) | 1 (1)
Discomfort at injection site when touched (General disorders) | 1 (1)
Patient felt faint (General disorders) | 1 (1)
Bilateral ear infection (Infections and infestations) | 1 (1)
Chest infection (Infections and infestations) | 1 (1)
Common cold (Infections and infestations) | 3 (4)
Patient visited the dentist and had a filling (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 9 (92)
Fall (Injury, poisoning and procedural complications) | 5 (9)
Bruising to right hip from fall (Injury, poisoning and procedural complications) | 1 (1)
Bruising to right shoulder following fall (Injury, poisoning and procedural complications) | 1 (1)
Bruising to the face following fall (Injury, poisoning and procedural complications) | 1 (1)
Fall up the stairs leading to flat due to increasing leg weakness (Injury, poisoning and procedural complications) | 1 (1)
Fall while getting out of bed, due to increase in leg weakness (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (6)
Blood bilirubin increased (Investigations) | 1 (4)
Cholesterol high (Investigations) | 5 (8)
Hemoglobin increased (Investigations) | 1 (1)
Abnormal CRP blood results (Investigations) | 1 (1)
Abnormal eosinophil blood results (Investigations) | 1 (1)
Abnormal glucose levels (3.1, normal results 3.5-11.0) (Investigations) | 1 (1)
Abnormal hdl level, clinically insignificant. (Investigations) | 1 (1)
Abnormal mean cell haemoglobin level, clinically insignificant (Investigations) | 1 (1)
Abnormal platelet distribution width result (Investigations) | 1 (1)
Abnormal ptt blood result (elevated) (Investigations) | 1 (1)
Abnormal red cell distribution levels (Investigations) | 1 (1)
Creatinine level decreased (Investigations) | 1 (1)
CRP increased (Investigations) | 1 (1)
Decreased aptt result (Investigations) | 1 (1)
Decreased basophil count (Investigations) | 1 (1)
Decreased basophil level (Investigations) | 2 (2)
Decreased basophil result (Investigations) | 4 (4)
Decreased creatinine (Investigations) | 1 (1)
Decreased creatinine levels (Investigations) | 1 (2)
Decreased creatinine result (Investigations) | 1 (1)
Decreased creatinine value - not clinically significant (Investigations) | 1 (1)
Decreased haematocrit value - not clinically significant (Investigations) | 1 (1)
Decreased haemoglobin value (Investigations) | 1 (1)
Decreased hdl cholesterol result (Investigations) | 2 (2)
Decreased hdl cholesterol value - not clinically significant (Investigations) | 1 (1)
Decreased hdl cholesterol value -not clinically significant (Investigations) | 1 (1)
Decreased hdl value - not clinically significant (Investigations) | 1 (1)
Decreased igm result (Investigations) | 1 (1)
Decreased monocyte result (Investigations) | 1 (1)
Decreased potassium level (Investigations) | 1 (1)
Decreased rbc dist width (Investigations) | 1 (1)
Decreased rbc distribution width (Investigations) | 2 (2)
Decreased red blood cell value - not clinically significant (Investigations) | 1 (1)
Decreased sodium levels (Investigations) | 1 (1)
Elevated aptt ratio (Investigations) | 1 (2)
Elevated ast blood level (Investigations) | 1 (1)
Elevated c- reactive protein blood results (Investigations) | 1 (1)
Elevated calcim level (Investigations) | 1 (1)
Elevated calcium level (Investigations) | 1 (1)
Elevated ck levels (Investigations) | 1 (1)
Elevated creatine kinase result (Investigations) | 1 (1)
Elevated crp result (Investigations) | 1 (1)
Elevated crp value - not clinically significant (Investigations) | 1 (1)
Elevated eosinophil result (Investigations) | 1 (1)
Elevated haematocrit blood level (Investigations) | 1 (1)
Elevated hdl cholesterol blood levels (Investigations) | 1 (1)
Elevated mean cell haemoglobin (Investigations) | 1 (1)
Elevated mean cell hb concentration (Investigations) | 1 (1)
Elevated mean cell hb level (Investigations) | 1 (1)
Elevated mean cell hb result (Investigations) | 2 (2)
Elevated monocyte result (Investigations) | 1 (1)
Elevated red blood cell count (Investigations) | 3 (4)
Elevated sodium levels (Investigations) | 1 (1)
Elevated total protein result (Investigations) | 1 (1)
Hdl cholesterol levels high (Investigations) | 1 (1)
Increased ck value - not clinically significant (Investigations) | 1 (1)
Increased crp level (Investigations) | 1 (1)
Increased eosinophils count - not clinically significant (Investigations) | 1 (1)
Increased esr value - not clinically significant (Investigations) | 1 (1)
Increased iga value - not clinically significant (Investigations) | 1 (1)
Increased monocyte count - not clinically significant (Investigations) | 1 (1)
Increased neutrophil count - not clinically significant (Investigations) | 1 (2)
Increased platelet dist width (Investigations) | 1 (1)
Increased platelet dist. width (Investigations) | 1 (1)
Increased rbc distribution width (Investigations) | 1 (1)
Increased white blood cell value - not clinically significant (Investigations) | 1 (1)
Low albumin level (Investigations) | 1 (1)
Low haematocrit (Investigations) | 1 (1)
Low sodium (Investigations) | 1 (1)
Mean cell hb concentration level elevated (Investigations) | 1 (1)
Prolonged pr interval on ecg (Investigations) | 1 (1)
Raised ast blood levels (Investigations) | 1 (2)
Raised ast levels (Investigations) | 1 (1)
Raised blood glucose level (Investigations) | 1 (1)
Raised crp result (Investigations) | 1 (1)
Raised eosinophil count (Investigations) | 1 (1)
Raised eosinophils (Investigations) | 1 (1)
Raised hdl cholesterol blood levels (Investigations) | 1 (1)
Raised sodium level (Investigations) | 1 (1)
Raised total protein result (Investigations) | 1 (1)
Reduced aptt ratio value - not clinically significant (Investigations) | 1 (1)
Reduced basophil count (Investigations) | 1 (1)
Reduced free thyroxine levels (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fractured nasal bone following fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased leg weakness leading to inability to stand resulting in admission to hospital (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasm in legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Occasional spasm in neck when yawning (Musculoskeletal and connective tissue disorders) | 1 (1)
Painful left shoulder blade (Musculoskeletal and connective tissue disorders) | 1 (1)
Right hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash on abdomen around injection site (Skin and subcutaneous tissue disorders) | 1 (1)
Rash on both feet (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to the COVID-19 pandemic, the high-risk status of trial patients, and the frequent hospital based visits, meant that both recruitment to the trial and further treatment was suspended after 11 patients had been recruited. As a result, patients were treated with interrupted and varying numbers of weekly ILB® treatments.

The pharmacokinetic evaluation was limited due to rejection of some poor quality blood samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Centre shall not publish or otherwise disseminate the conclusions of the Study, including all or any part of the Results of the Study without the prior written consent of the Sponsor, such consent not to be unreasonably withheld or delayed. Any publication or other dissemination of the conclusions of the Study by the National Health Organisation (NHS) Organisation shall not' occur until the Sponsor has published the conclusions of the Study.

Results published- PubMed ID: 38990927

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT03705390/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT03705390/SAP_001.pdf